CLINICAL TRIAL: NCT02981199
Title: A Prospective, Multi-center, Randomized Controlled Trial of Microtransplantation Versus Auto-SCT in ≥PR Multiple Myeloma Patients
Brief Title: Microtransplantation Versus Auto-SCT in ≥PR Multiple Myeloma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Wenming (Other)
Collaborators: 307 Hospital of PLA (Other)
Responsible Party: Sponsor-Investigator, Chen Wenming, professor, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-MSCT-001
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Microtransplantation; Autologous Stem Cell Transplantation; Multiple Myeloma in Relapse
Keywords: microtransplantation; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Stem Cell Transplantation

ARMS (2):
- Micro-SCT (Active Comparator): patients treated with microtransplantation. [VMD chemotherapy(bortezomib 1.3mg/m2 d1,4,8,11; melphalan 60mg/m2 d1; dexamethasone 20mg d1,2,4,5,8,9,11,12) + low dose allogeneic stem cell transplantation]×4cycles; [PTD chemotherapy(bortezomib 1.3mg/m2 d1,4,8,11; thalidomide 100mg/d, dexamethasone 20mg d1,2,4,5,8,9,11,12)]×1cycle; then maintenance therapy with thalidomide 100mg/d.
  microtransplantation = [VMD regimen chemotherapy+ low dose allogeneic stem cell transplantation]×4cycles
  Interventions: Procedure: stem cell transplantation
- Auto-SCT (Active Comparator): patients treated with Auto-SCT. conditioning with Mel+Vel regimen (melphalan 200mg/m2 d-2, bortezomib 1.3mg/m2 d-6,-3,+1,+4) + autogeneic stem cell transplantation; [PTD chemotherapy(bortezomib 1.3mg/m2 d1,4,8,11; thalidomide 100mg/d, dexamethasone 20mg d1,2,4,5,8,9,11,12)]×4cycle; then maintenance therapy with thalidomide 100mg/d.
  Interventions: Procedure: stem cell transplantation

INTERVENTIONS:
Procedure: stem cell transplantation — conditioning with chemotherapy [VMD regimen(bortezomib, melphalan, dexamethasone) or Mel+Vel regimen(melphalan, bortezomib)], then stem cell transfusion

SUMMARY:
Comparison of the efficacy and safety of microtransplantation and autologous transplantation in the treatment of ≥PR multiple myeloma patients, 2-year PFS and OS were also been observed. To identify the role of microtransplantation in the treatment of multiple myeloma.

DETAILED DESCRIPTION:
NDMM patients induction therapy with 4 cycles PCD/PAD regimen, achieve ≥PR, eligible for SCT, were randomly divided into two arms. One arm receive microtransplantation, and the other accept auto-SCT. Comparison of the efficacy and safety of two arms, 2-year PFS and OS were also been observed. Clear the above program related hematopoietic recovery, remission rate, infection and recurrence rate, survival rate and the formation of micro inlay, minimal residual disease and GVHD, etc. To identify the role of microtransplantation in the treatment of multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis MM compliance with IMWG diagnostic criteria(2014)
2. induction therapy with 4 cycles PCD/PAD regimen, achieve ≥PR
3. KPS ≥60，ECOG≤2 4）Age 18-65，eligible for SCT 5）Heart function < II level (NYHA standard) and ejection fraction > 50% -

Exclusion Criteria:

1. KPS<60
2. Allergy to bortezomib,epirubicin, or drug ingredients
3. Severe hepatitis and organ dysfunction: a serious infection has not been controlled; cardiac ejection fraction <50%, serum bilirubin >3mg/dl, severe abnormal results of liver function test (AST is greater than 3 times the upper limit), severe renal injury; central nervous system disorders, uncontrolled mental illness
4. With more than 2 bortezomib associated with peripheral neuropathy or neuralgia patients
5. Patients with active stage of the herpes zoster
6. Women in pregnancy or lactation
7. MM with AL or EM plasma cell tumor
8. The patient refused to accept the above treatment and signature
9. Donor does not meet the requirements: including HIV positive, active hepatitis B, bone marrow disease, donor refused to provide hematopoietic stem cells and do not agree to sign.
10. Epirubicin / other anthracyclines previously accumulated more than 240mg/m2 -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years
overall survival | 2 years

SECONDARY OUTCOMES:
rate of complete remission | 2 year
minimal residual disease | 2 year
hematopoietic recovery | 3 month
infection | 3 month
GVHD | 1 year
relapse | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Chen, doctor, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No